CLINICAL TRIAL: NCT02423759
Title: A Randomized Controlled Trial Comparing Rectal Swab Culture Based Chemoprophylaxis Versus Combined Single-Shot Gentamycin and Ciprofloxacin Versus Ciprofloxacin Alone for Peri-procedure Chemoprophylaxis During Transrectal Prostate Biopsy.
Brief Title: A Trial Assessing Peri-procedure Chemoprophylaxis During Transrectal Prostate Needle Biopsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Elshal, Dr, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MANS-2015-03
Record Dates: First submitted 2015-03-24; First posted 2015-04-22 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Benign Prostate Hyperplasia
Keywords: Chemoprevention
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Ciprofloxacin; Gentamicins

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- ciprofloxacin (Active Comparator): standard chemoprophylaxis [500mg ciprofloxacin twice daily for 3 days]
  Interventions: Drug: ciprofloxacin
- ciprofloxacin and gentamycine (Experimental): Augmented Chemoprophylaxis [standard chemoprophylaxis plus 160mg]
  Interventions: Drug: ciprofloxacin and gentamycine
- culture based chemoprophylaxis (Experimental): Patients will receive antibiotic according to rectal swab culture at time of biopsy and then after for 3 days.
  Interventions: Drug: culture based chemoprophylaxis

INTERVENTIONS:
Drug: ciprofloxacin — 500mg ciprofloxacin twice daily starting the day before biopsy and continued for 3 days after
  Other Names: standard chemoprophylaxis
  Arms: ciprofloxacin
Drug: ciprofloxacin and gentamycine — standard chemoprophylaxis plus gentamicin 160mg intramuscular once just before the biopsy
  Other Names: standard chemoprophylaxis plus gentamicin
  Arms: ciprofloxacin and gentamycine
Drug: culture based chemoprophylaxis — Patients will receive antibiotic according to rectal swab culture at time of biopsy and then after for 3 days.
  Arms: culture based chemoprophylaxis

SUMMARY:
The aim of the study is to evaluate whether changing antibiotic prophylaxis from fluoroquinolones alone to fluoroquinolones plus gentamicin 160mg single IM dose or targeted antibiotic prophylaxis according to rectal swab culture would influence infectious complication rates in those men undergoing transrectal ultrasound-guided prostate biopsy.

DETAILED DESCRIPTION:
Introduction Transrectal ultrasound (TRUS) guided prostate biopsy is the standard procedure for the histological diagnosis and grading of prostate cancer that consequently help in providing the appropriate line of treatment. Risks of infectious complications post TRUS-guided biopsy have increased in the last years.

In their study, a total of 5798 TRUS-guided biopsies performed between 2002 and 2011. Increased incidence of infectious complications is noted from 0.52 infections per 100 biopsies between 2002 and 2009 to 2.15 infections per 100 biopsies between 2010 and 2011 (P< 0.001). The commonest organism found to be responsible for these infectious complications is Escherichia coli (E. Coli).

The American Urological Association best practice policy statement recommends antibiotic prophylaxis prior to transrectal prostate biopsy. The current practice is to give patients a dose of an oral fluoroquinolone (FQ) 30 to 60 minutes before biopsy and to be continued for 2 to 3 days after.

Recent studies show that 2% of patients will develop febrile urinary tract infection or even urosepsis and require hospitalization for intravenous antibiotics . There is considerable concern regarding the rising incidence of community-acquired antibiotic-resistant organisms.

It is proposed that resistant organisms are introduced into the bladder and the blood stream from the rectum during the procedure that's why patients already colonized with these resistant organisms may be at higher risk. Thereby, some authors suggest a targeted rectal swab culture before (TRUS)-guided biopsy then giving the appropriate antibiotic prophylaxis aiming at reducing post biopsy infection rates while minimizing unnecessary broad-spectrum antibiotic use.

Retrospective data showed that septicemia was seen in 24 of 300 (8%) and 15 of 897 (1.7%) in patients receiving peri-procedure ciprofloxacin alone and patients receiving ciprofloxacin plus single IV dose of amikacin injection respectively (p=0.001). E. Coli resistant to quinolones was responsible for 33 of 39 (84.6%) septicemic cases. In a retrospective study in UK, 12.9% developed infectious complications following prostate biopsy in patients receiving co-amoxiclav and gentamycin.

In another retrospective study, hospitalization rate due to post-biopsy infections was 3.8% compared to 0.6% (p=0.001) in patients receiving the standard ciprofloxacin and augmented prophylaxis with ciprofloxacin plus single IM 80mg gentamycin respectively. Of the admitted patients who received standard prophylaxis, 73% had fluoroquinolone resistant E. Coli urinary infection and/or bacteremia and only 9% had strains resistant to gentamicin. Multivariate analysis showed that the standard regimen was significantly associated with hospital admission due to post-biopsy infection. The augmented regimen resulted in a cost savings of $15,700 per 100 patients compared to the standard regimen.

Diabetes was found in 4% of the fluoroquinolone sensitive group vs 14.7% of the resistant group (p < 0.001). Biopsy history was not associated with resistance.

Urosepsis is a systemic reaction of the body to a bacterial infection of the urogenital organs with the risk of life-threatening events including shock. Systemic inflammatory response syndrome (SIRS) criteria are defined as 2 or more of the following variables; increase in body temperature to 38°C or more, heart rate of more than 90 beats per minute, respiratory rate of more than 20 per minute or arterial carbon dioxide tension (PaCO2) less than 32mm Hg and abnormal white blood cell count (>12,000/µL or < 4,000/µL) Aim of the work; The aim of the study is to evaluate whether changing antibiotic prophylaxis from fluoroquinolones alone to fluoroquinolones plus gentamicin 160mg single IM dose or targeted antibiotic prophylaxis according to rectal swab culture would influence infectious complication rates in those men undergoing transrectal ultrasound-guided prostate biopsy.

ELIGIBILITY:
Inclusion Criteria:

1. Prothrombin concentration > 70%
2. Platelet count > 100.000/cm

Exclusion Criteria:

1. Acute prostatitis (positive symptoms and signs)
2. Patients with compromised renal function (serum creatinine >1.6 mg/dl)
3. Uncontrolled DM
4. Patients on immunosuppressive therapy
5. Active steroid intake
6. Untreated bleeding diathesis

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 510 (Actual)
Dates: Start 2015-04; Primary Completion 2017-01-16 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
occurrence of post procedure infectious complications | 2 weeks
  occurrence of post procedure infectious complications (e.g urosepsis and local genital or prostate infectious complications). Sepsis is identified as occurrence of two or more of SIRS criteria.

SECONDARY OUTCOMES:
flouroquinolones resistance in rectal carriage | 2 weeks
  identification of the prevalence of flouroquinolones resistance in rectal carriage in this subset of patients and post procedure non-infectious complications.
post procedure non-infectious complications | 2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Elshal, MD, Principal Investigator — Mansoura University
Locations (1):
- Urology and Nprhology Center, Al Mansurah, Aldakahlia, Egypt